CLINICAL TRIAL: NCT01625065
Title: Toxicological Analyses of Blood and Urine Samples in Pain Patients and Pre-surgical Control Patients to Investigate Incidences of Concealed and Feigned Substances
Brief Title: Study of Medication Compliance - a Comparison of Patients in Pain Management and Pre-surgical Patients
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr. med., Ruhr University of Bochum
Other Study IDs: Medi-3889-10
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Pain
Keywords: medication compliance; adherence; toxicological analyzes; GC-MS; HPLC; pain patients; opioid misuse; patients with current pain
MeSH Terms: conditions — Pain; Medication Adherence; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pain patients: patients from a specific pain management department, patients with long duration of pain, mostly insufficiently treated pain
- pre-surgical patients: patients from a surgical outpatient department with current pain

SUMMARY:
In this study medication compliance regarding current drug use is investigated using toxicological analyzes in two patient groups: patients from a pain management department and pre-surgical control patients. The aim is to explore the incidence of concealed and feigned substances and to determine the respective substance classes. Expecting that noncompliance is higher in the pain patient group, the investigators want to identify clinical risk factors for noncompliant drug report.

ELIGIBILITY:
Inclusion Criteria:

* provided informed consent
* current pain

Exclusion Criteria:

* no taking of blood sample possible
* no consent with toxicological analyzes
* insufficient comprehension of the German language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pain management and surgical outpatient department of a University hospital
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Bergmannsheil, Bochum, Germany

REFERENCES:
- [Derived] Kipping K, Maier C, Bussemas HH, Schwarzer A. Medication compliance in patients with chronic pain. Pain Physician. 2014 Jan-Feb;17(1):81-94. PMID 24452648